CLINICAL TRIAL: NCT02087449
Title: A Prospective Multi-center Study on E1 Acetabular Liner in THA
Brief Title: Evaluate E1 Wear, Clinical Performance of E1 Liner in THA in Korean Patient Population
Acronym: E1Hip
Status: Terminated | Type: Observational
Why Stopped: Sponsor decided to terminate study.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: INT.CR.GH5.13
Record Dates: First submitted 2014-03-05; First posted 2014-03-14 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis; Avascular Necrosis; Traumatic Arthritis; Rheumatoid Arthritis; Legg-perthes Disease
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Legg-Calve-Perthes Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- E1-Hip Bearing: E1-Hip Bearing, Evaluate E1 Wear, Clinical Performance of E1 Liner in THA in Korean Patient Population
  Interventions: Device: E1-Hip Bearing

INTERVENTIONS:
Device: E1-Hip Bearing — Vitamin E doping of highly cross-linked polyethylene is a proposed method for insuring long-term oxidative stability of highly cross-linked ultra-high molecular weight polyethylene for use in total joint arthroplasty. In vitro research and development studies have shown that this material has improved wear performance, retention of mechanical properties, and a high resistance to oxidation due to the anti-oxidative properties of Vitamin E.

SUMMARY:
Evaluate E1 wear, Clinical Performance of E1 liner in THA in Korean Patient Population

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is one of the most successful surgical procedures in general. Yet, a few problems remain unsolved, and aseptic loosening is probably the most important of them. One of the main reasons for aseptic loosening in THA is the foreign body reaction caused by the wear particles. Since the late 1990s, the orthopedic industry has been developing highly crosslinked polyethylene (HXLPE) materials to capitalize on the increased wear resistance. In 2007, E1® Antioxidant Infused Technology was developed to reduce wear rate, maintain mechanical properties and prevent oxidative degradation.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in this study if they received Ringloc acetabular system with E1 liner per the approved indications for use by KFDA in Korea. Specifically,

1. Osteoarthritis
2. Avascular necrosis
3. Legg Perthes
4. Rheumatoid Arthritis
5. Diastrophic variant
6. Fracture of the pelvis
7. Fused hip
8. Slipped capital epiphysis
9. Subcapital fractures
10. Traumatic arthritis Patients aged over 20 Patients with limited co-morbidity - ASA I - III

Exclusion Criteria:

Exclusion Criteria for this study should comply with the stated contraindications on package inserts of Ringloc acetabular system with E1 liner. These indications are stated below:

Absolute contraindications include: infection, sepsis, and osteomyelitis

Relative contraindications include:

1. uncooperative patient or patient with neurologic disorders who are incapable of following directions,
2. osteoporosis,
3. metabolic disorders which may impair bone formation,
4. osteomalacia,
5. distant foci of infections which may spread to the implant site,
6. rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram, and
7. vascular insufficiency, muscular atrophy, or neuromuscular disease.
8. pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated to have Total Hip Arthroplasty at Daegu Catholic University Hospital, Kyung Pook Nat'l Univ. Hospital, Yeonsei Univ. College of Medicine, and Gangdong Kyung Hee Univ. Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
HHS score | 1 year
  Comparison in clinical outcomes scores between preoperative and various postoperative time points

SECONDARY OUTCOMES:
Hip Functions | 6 Months
  Harris Hip Score at post follow-up visit
EQ5D | 6 Months
  Standardised instrument for use as a measure of health outcome
Modified University of California Los Angeles (UCLA) Activity Score | 6 Months
  It asks patients to rate their activity level from 1 to 10, with 1 defined as "no physical activity" and 10 defined as "regular participation in impact sports".
  The UCLA scale has demonstrated construct validity, excellent reliability, and the best completion rates.
Radiographic Assessment | Immediate post-op(2 - 4 Weeks)
  Radiographic Assessment at Immediate post-op(2 - 4 Weeks), 6 months, 1 year, 2 year, 5 year postop
Hip Functions | 1 year
  Harris Hip Score at post follow-up visit
Hip Functions | 2 years
  Harris Hip Score at post follow-up visit
Hip Functions | 5 years
  Harris Hip Score at post follow-up visit
EQ5D | 1 year
  Standardised instrument for use as a measure of health outcome
EQ5D | 2 years
  Standardised instrument for use as a measure of health outcome
EQ5D | 5 years
  Standardised instrument for use as a measure of health outcome
Modified University of California Los Angeles (UCLA) Activity Score | 1 year
  It asks patients to rate their activity level from 1 to 10, with 1 defined as "no physical activity" and 10 defined as "regular participation in impact sports".
  The UCLA scale has demonstrated construct validity, excellent reliability, and the best completion rates.
Modified University of California Los Angeles (UCLA) Activity Score | 2 years
  It asks patients to rate their activity level from 1 to 10, with 1 defined as "no physical activity" and 10 defined as "regular participation in impact sports".
  The UCLA scale has demonstrated construct validity, excellent reliability, and the best completion rates.
Modified University of California Los Angeles (UCLA) Activity Score | 5 years
  It asks patients to rate their activity level from 1 to 10, with 1 defined as "no physical activity" and 10 defined as "regular participation in impact sports".
  The UCLA scale has demonstrated construct validity, excellent reliability, and the best completion rates.
Radiographic Assessment | 6 Months
  Radiographic Assessment at Immediate post-op(2 - 4 Weeks), 6 months, 1 year, 2 year, 5 year postop
Radiographic Assessment | 1 year
  Radiographic Assessment at Immediate post-op(2 - 4 Weeks), 6 months, 1 year, 2 year, 5 year postop
Radiographic Assessment | 2 years
  Radiographic Assessment at Immediate post-op(2 - 4 Weeks), 6 months, 1 year, 2 year, 5 year postop
Radiographic Assessment | 5 years
  Radiographic Assessment at Immediate post-op(2 - 4 Weeks), 6 months, 1 year, 2 year, 5 year postop

CONTACTS AND LOCATIONS:
Overall Officials: Shin Yoon Kim, PHD, Principal Investigator — Kyung Pook Nat'l Univ. Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, Kyungsangbuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT02087449/Prot_SAP_000.pdf